CLINICAL TRIAL: NCT00218946
Title: Nasogastric Tube in Premature Babies - Pain and Treatment. A Randomised, Partly Blinded, Placebo-controlled Factorial Clinical Trial of Sucrose and Pacifier
Brief Title: Nasogastric Tube in Premature Babies - Pain and Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: NISE-2005-1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Infant, Premature
Keywords: pain; infant, premature; intubation, gastrointestinal; Neonatal nursing
MeSH Terms: conditions — Premature Birth; Pain | interventions — Sucrose; Pacifiers

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- control (No Intervention): no fluid, no pacifier
- water (Experimental): water, no pacifier
  Interventions: Other: sterile water
- sucrose (Experimental): Sucrose, no pacifier
  Interventions: Drug: Sucrose
- pacifier (Experimental): No fluid, pacifier
  Interventions: Device: Pacifier
- water and pacifier (Experimental): water, pacifier
  Interventions: Device: Pacifier
- sucrose and pacifier (Experimental): sucrose, pacifier
  Interventions: Drug: Sucrose; Device: Pacifier

INTERVENTIONS:
Drug: Sucrose — 30 % sucrose
  Arms: sucrose; sucrose and pacifier
Device: Pacifier
  Arms: pacifier; sucrose and pacifier; water and pacifier
Other: sterile water
  Arms: water

SUMMARY:
Does sucrose or pacifier influence pain in premature babies when a nasogastric tube is inserted?

DETAILED DESCRIPTION:
A total of 24 premature babies are randomised to receive either placebo (sterile water), 30 % sucrose, or pacifier in a complete factorial, cross-over design. Pain is rated on the PIPP scale by observers blinded to the procedure other than use of pacifier.

ELIGIBILITY:
Inclusion Criteria:

* 28 - 32 weeks gestational weeks
* not on mechanical ventilation

Exclusion Criteria:

* high risk group regarding cerebral prognosis

Ages: 3 Days to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pain measured on PIPP (Premature Infant Pain Profile) scale | 4 week to complete

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Skogvoll, MD, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- St. Olavs University Hospital, Trondheim, Trondheim, Norway

REFERENCES:
- [Background] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730
- [Result] Kristoffersen L, Skogvoll E, Hafstrom M. Pain reduction on insertion of a feeding tube in preterm infants: a randomized controlled trial. Pediatrics. 2011 Jun;127(6):e1449-54. doi: 10.1542/peds.2010-3438. Epub 2011 May 2. PMID 21536607